CLINICAL TRIAL: NCT01058278
Title: Impact of the Post-operative Treatment on the Intraocular Pressure Post Selective Laser Trabeculoplasty (SLT) on Patients With Primary Open-angle Glaucoma
Brief Title: Impact Post-operative Treatment on Intraocular Pressure Post-SLT on Patients With Primary Open-angle Glaucoma
Acronym: SLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Glaucoma Clinical Research Council (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Béatrice Des Marchais, Chercheure clinicienne associée, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DR-002-1213
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Glaucoma; Inflammatory Response
Keywords: Glaucoma; Ocular Hypertension; Intraocular Pressure; Trabeculectomy
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prednisone acetate 1% (Active Comparator): A topic cortisone-based treatment
  Interventions: Procedure: Selective Laser trabeculoplasty
- diclofenac 0.1% (Active Comparator): an non-steroidal anti-inflammatory drug
  Interventions: Procedure: Selective Laser trabeculoplasty
- Artificial Tears (Placebo Comparator): Pharmasciences DIN: 02229570
  Interventions: Procedure: Selective Laser trabeculoplasty

INTERVENTIONS:
Procedure: Selective Laser trabeculoplasty — The Selective Laser Trabeculoplasty is done with the Latina lens after applying a drop of iopidine in the treated eye and alcaïne in both eye. Fifty spots are done over 180°. The maximal and total energy is written in the chart. After the treatment, prednisolone acetate 1% (a corticosteroid), diclofenac 0.1% (an NSAID) or a placebo is used. The three treatments were administered 4 times a day (at breakfast, lunch, dinner and at bedtime) for five days.

SUMMARY:
The present study's main objective is to assess if there is a significant difference between either of the treatments frequently used in post-op, namely a topic cortisone-based treatment, an non-steroidal anti-inflammatory drug (NSAID) or simply a placebo, in order to gain the best long term (6 months) efficacy of the SLT.

DETAILED DESCRIPTION:
The selective laser trabeculoplasty (SLT) is the laser treatment of choice for treating glaucoma. A There is however a controversy regarding the use of drops post-treatment. Indeed, some would prefer not to pharmacologically modulate the post-op inflammatory response which can be an integral part of the treatment by favouring the mobilisation of the macrophages which participate to the trabeculae "cleaning". Others will prefer to calm the inflammatory reaction and choose an anti-inflammatory drug (either steroidal or non-steroidal).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from with primary open-angle glaucoma.
* Patients with IOP > 21 mmHg, uncontrolled with medical treatment or due to non-compliance, or to whom this is the first glaucoma treatment.
* Patients > 18 years old, able to consent.
* Patients consenting to the trial.

Exclusion Criteria:

* Patients suffering from chronic glaucoma other than primary open-angle glaucoma
* Patients who had changes done to their anti-glaucoma treatments over the last 6 weeks or following the SLT
* Patients under oral corticosteroid treatment at the time of the operation or those who have stopped during the preceding month.
* Patients suffering from an important corneal disease which interferes with the capacity to visualize the entire trabeculae.
* Monophthalmic patients.
* Patients who already underwent a glaucoma treatment to the eye requiring treatment.
* Patients who already underwent a glaucoma treatment using SLT or ALT (Argon laser trabeculoplasty)
* Patients who underwent cataract surgery in the past 3 months.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure in the treated eye | 1 hour, 7 days, 1.5, 3 and 6 months

SECONDARY OUTCOMES:
Side effects (include a slight uveitis, oculary discomfort and a spike in intraocular pressure in the immediate post-op period) | 1 hour, 7 days, 1.5 months, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice Des Marchais, FRCSC M.Sc., Principal Investigator — CHU de Quebec-Universite Laval
Locations (1):
- Centre universitaire d'ophtalmologie, Hôpital du Saint-Sacrement, CHU de Québec, Québec, Quebec, Canada